CLINICAL TRIAL: NCT02485743
Title: A Randomized, Double-blind Multi-centre Trial Comparing a Diet Including Satiating Products Compared to Control Products - SATIN Satiety Diet - Proof of Concept
Brief Title: A Trial Comparing a Diet Including Products Aimed at Targeting Satiety
Acronym: SATIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Jason Halford (Other)
Collaborators: University of Copenhagen (Other); University Rovira i Virgili (Other)
Responsible Party: Sponsor-Investigator, Professor Jason Halford, Professor Jason Halford, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NEXS-B292
Record Dates: First submitted 2015-06-25; First posted 2015-06-30 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Weight; Appetite
Keywords: satiation; satiety; weight loss; maintained weight loss
MeSH Terms: conditions — Body Weight; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Diet Products (Active Comparator): A range of products that will be provided as part of a weight maintenance diet which contain active ingredients aimed at increasing satiety (such as inulin, β-glucan, protein and mycoprotein). All ingredients are accepted food ingredients approved for human consumption in Europe.
  Interventions: Other: Active Diet Products
- Placebo Diet Products (Placebo Comparator): A range of products matching those provided in the Active Diet which will be provided as part of a weight maintenance diet but do not contain additional ingredients aimed at improving satiety (food matrices will be the same - e.g. shakes, cheeses etc but without active ingredients).
  Interventions: Other: Placebo Diet Products

INTERVENTIONS:
Other: Active Diet Products — A range of Active Diet Products that will be provided as part of a weight maintenance diet which contain active ingredients aimed at increasing satiety (such as inulin, β-glucan, protein, and mycoprotein). All ingredients are accepted food ingredients approved for human consumption in Europe.
  Arms: Active Diet Products
Other: Placebo Diet Products — A range of Placebo Diet Products matching those provided in the Active Diet which will be provided as part of a weight maintenance diet but do not contain additional ingredients aimed at improving satiety (food matrices will be the same - e.g. shakes, cheeses etc but without active ingredients).
  Arms: Placebo Diet Products

SUMMARY:
This multi-centre, randomised controlled trial will be conducted over 12-weeks to evaluate whether lower appetite is associated with weight loss maintenance success. The effect of a healthy diet supplemented with products that could enhance feelings of satiety and reduce food intake after an initial weight loss period to assess weight maintenance. Participants will either receive the active SATIN product or a matched control product. The products contain ingredients which have been shown to positively affect satiety, satiation and/or body weight and are all accepted food ingredients approved for human consumption in Europe. They will be incorporated into different food matrices, e.g. drinks, shakes and cheeses. Corresponding control products without the active ingredients will be provided to participants allocated to the control group. The participants will be instructed in detail on how and when to consume the test products. Participants will be 300 adults (BMI >27kg/m2; Age>18years) who will be tested at three research sites (University of Liverpool, United Kingdom; University of Copenhagen, Denmark and University Rovira I Virgili, Spain). Recruitment will be divided between sites. Participants will attend assessments at one of the three research sites continually throughout the study period. The primary outcome is to assess potential associations between changes in appetite (ad libitum energy intake, acute as well as sustained) and change in body weight during the 12-week follow-up period. Secondary outcomes include assessing waist circumference, body composition (DXA), subjective appetite, biomarkers of health outcomes (blood and urine indices), changes in physical activity as well as consumer benefits of the trial (assessed in a range of questionnaires) to determine diet efficacy.

DETAILED DESCRIPTION:
The study is a double blinded parallel randomized multicentre study, with six arms. The study will be conducted simultaneously in Denmark, Spain and United Kingdom, at the study sites specified on page 3. A total of 300 participants with an initial BMI of 27 to 35 kg/m2 and a fat mass of no less than 23% will be enrolled in the study. An initial weight loss of a minimum of 8 % will be needed for inclusion in the randomized part of the study. The weight loss will be achieved by administration of a low calorie diet (LCD) for 8 weeks managed by dietician supervised group sessions. Failure to reach at least 8% weight reduction during the LCD will result in exclusion from the intervention.

Participants reaching the pre-defined weight loss of no less than 8% will enter a 7-10 days run-in period for diet stabilization before entering the 12-week randomized part of the study. In the randomized part of the study all participants will be advised to follow a general healthy weight loss maintenance diet in accordance with national dietary guidelines. In addition, participants will be randomly allocated in a 1:1 ratio to one of the following intervention groups; 1) including an active satiety enhancing product (active intervention group) or 2) including a similar control product without satiety enhancing properties (control group).

For both groups, the participants will be instructed to consume the intervention products daily. Primary study visits for the assessment of body weight, waist circumference, hip circumference, sagittal diameter and blood pressure will be performed at the beginning, and at the end of the intervention period. At least every four weeks during the intervention, the participants will be requested to pick up the study products, and during these visits bodyweight and waist and hip circumference will be recorded. The participants will furthermore meet individually with a dietician three times during the 12 weeks intervention period to enhance compliance with the weight loss maintenance diet and to ensure incorporation of the study specific products into their diet as instructed. Adverse events and concomitant medicine will be registered continuously throughout the study. For each participant, the total study duration is 24 weeks, and includes 17 visits at the study site in total (14+3 appetite probe days)

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27,0 and ≤ 35,0 kg/m2
* Fat mass ≥ 23 % as assessed by bio impedance at the screening visit
* Healthy
* Acceptance of the experimental foods
* Provided voluntary written informed consent

Exclusion Criteria:

* < 8.0% weight loss during the Low Calorie Diet (LCD) period (will be assessed at visit 7 after having completed the 8 week LCD period)
* Dislike ≥ 25% of the study products (will be assessed at visit 7 through test tasting)
* Known diseases which may affect energy expenditure and/or satiation/satiety/food intake i.e. inflammatory bowel disease, thyroid deceases, major depressions and bipolar deceases
* Eating behaviour characteristics (e.g. restrained eating, disinhibition, emotional eating) identified at the screening visit based on questionnaires
* Weight changes ±3 kg in the last three months
* Dietary patterns interfering with the study protocol, as judged by the Investigator (e.g. vegetarian, vegan, low carb dieters, high fat dieters) two months prior inclusion, during the study or plans to initiate during the study
* Severe food allergies and food intolerances expected to interfere with the study
* Engagement in elite sports or similar strenuous exercise ≥ 5h/week
* Pregnancy or lactation, pregnancy within the past 12 month or plans to become pregnant during the study
* Smoking, smoking cessation within the past three months and/or nicotine use (including electronic cigarettes)
* Medical conditions as known by the participants:

  * Diabetes mellitus (type 1 and 2) (History of gestational diabetes mellitus is allowed)
  * Cardiovascular disease including current angina; myocardial infarction; coronary revascularization procedures; stroke (either ischemic or hemorrhagic, including transient ischemic attacks); symptomatic peripheral artery disease that required surgery or was diagnosed with vascular imaging techniques; ventricular arrhythmia; uncontrolled atrial fibrillation; congestive heart failure (New York Heart Association Class II or IV); hypertrophic myocardiopathy; and history of aortic aneurism ≥5.5 cm in diameter or aortic aneurism surgery within the past six months, as diagnosed by a medical doctor
  * Systolic blood pressure above 160 mmHg and/or diastolic blood pressure above 100 mmHg whether on or off treatment for hypertension. If being treated, stable treatment (i.e. no change in treatment, either dose, type of medication or other changes) within last 3 months is required
  * Chronic kidney disease defined as either kidney damage or estimated Glomerular Filtration Rate (eGFR) of less than 60 mL/min/1.73m2 or Creatinine >1.5 times upper limit of normal (according to local laboratory reference values) for longer than 3 months as diagnosed by a medical doctor
  * Liver disease e.g. cirrhosis (fatty liver disease allowed), or liver dysfunction with transaminases (Alanine Transaminase (ALT) and/or Aspartate Transaminase (ASAT)) more than 3 times the upper limit of normal (according to local laboratory reference values) as diagnosed by a medical doctor
  * Active inflammatory bowel disease, celiac disease, chronic pancreatitis or other disorder potentially causing malabsorption
  * Cancer - active malignant cancer or history of malignancy within the last 5 years (with exception of local basal and squamous cell skin cancer).
  * Previous bariatric surgery or intention to undergo bariatric surgery within the next 12 months
  * History of extensive small or large bowel resection
  * Known endocrine origin of obesity (except for treated hypothyroidism)
  * Transmissible blood-borne diseases e.g. hepatitis B, HIV
  * Any recent surgical procedure not fully recovered (as judged by the investigator)
* Current use of prescription medication or use within the previous month that has the potential of affecting body weight such as systemic corticosteroids (excluding inhaled and topical steroids) psychoactive medication, epileptic medication, or weight loss medications (either prescription, over the counter or herbal). Low dose antidepressants are allowed if they, in the judgment of the investigator, do not affect body weight or participation in the study protocol. Levothyroxine for treatment of hypothyroidism is allowed if the participant has been on a stable dose for at least 3 months
* Current use of prescription medication that does not affect body weight should have been stable for the past 3 months and expected to be stable during the study
* Concurrent therapy with immunosuppressive drugs or cytotoxic agents
* Haemoglobin concentration below local laboratory reference values (i.e. anaemia)
* Blood donation or transfusion within the past month before screening or during the study
* Regularly consumption of alcohol above recommendations; > 21 alcoholic units/week (men), or > 14 alcoholic units/week (women)
* Drug abuse, as judged by the investigator, within the previous 12 months
* Psychological or behavioural problems which, in the judgement of the investigator, would lead to difficulty in complying with the study protocol
* Psychiatric disorders: schizophrenia, bipolar disease, eating disorders, or depression with hospitalization within the last 6 months.
* Participation in other clinical trials within the past three months or intention to do so during the study, which are likely to affect the present study
* History of repeated failure to complete a LCD
* Allergy or intolerance for components of the LCD product
* Unable to follow the recommended diet for religious reasons, swallowing disorders, other physiological reasons or any other reasons for not being able to follow the recommended diet
* Inability or unwillingness to give written informed consent or communicate with study personnel
* Inability or unwillingness to follow the study protocol and instructions giving by the study personnel
* Institutionalization - permanent or long-stay resident in a care home or similar institution
* Illiteracy
* Any other condition that judged by the investigator may interfere with the adherence to the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in appetite related to change in maintained weight loss | First measured after the 8-week Low Calorie Diet period then over the 12-week intervention period
  * Δenergy intake between standard appetite probe day and random appetite probe day before initiating the intervention vs. Δbody weight before initiating the intervention and after completing the intervention (short term/acute effect on appetite) using data from all subjects (active and standard).
  * Δenergy intake between standard appetite probe day and random appetite probe day after initiating the intervention vs. Δbody weight before initiating the intervention and after completing the intervention (long term effect on appetite) using data from all subjects (active and standard).

SECONDARY OUTCOMES:
Change in subjective appetite related to change in maintained weight loss | : First measured after the 8-week Low Calorie Diet period then after the 12-week intervention period
  * Δcomposite subjective appetite ratings as well as Δsatiety and Δfullness ratings between standard appetite probe day and random appetite probe day before initiating the intervention vs. Δbody weight before initiating the intervention and after completing the intervention using data from all subjects (active and standard).
  * Δcomposite subjective appetite ratings or each of the appetite ratings between standard appetite probe day and random appetite probe day after initiating the intervention vs. Δbody weight before initiating the intervention and after completing the intervention (long term effect on appetite) using data from all subjects (active and standard).
  * Ratings of hunger, desire to eat as well as prospective food consumption at standard appetite probe day vs. Δbody weight before initiating the intervention and after completing the intervention
To test if subjects receiving the active products (enhanced satiating power) will have a better weight-maintenance compared to subjects receiving control products (standard products). This will be tested with the 3 products combined in the main study. | First measured after the 8-week Low Calorie Diet period then after the 12-week intervention period
  - Difference in weight-regain (Δbody weight before initiating the intervention and after completing the intervention) between active and control products.
Change in body composition | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Body composition will be assessed through dual X-ray absorptiometry (DEXA) scans at 3 points throughout the trial to assess changes in body composition as a consequence of the low calorie diet and the intervention diet
Biomarkers of appetite/metabolomics (Method: NMR; units; mM) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method: Nuclear magnetic resonance (NMR); Unit: mM; Variables: Free_Cholesterol, Esterified_Cholesterol, Total_Cholesterol, Triglycerides, Phosphatidylcholine, Lysophosphatidylcholine, Sphingomyelin
Biomarkers of appetite/metabolomics (Method: NMR; units: % of FA Chains) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = Nuclear Magnetic resonance (NMR); Units = % of FA chains; variables = fatty acyl chains, Omega 3 fatty acid, Arachidonic-eicosapentaenoic acid, docosahexaenoic acid, linoleic acid, polyunsaturated fatty acids, monounsaturdated fatty acids.
Biomarkers of appetite/metabolomics (Method: LC; units: mM; part 1) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = Liquid Chromatography (LC); Units = mM; variables = C14.0 LPC (lysophosphatidylcholine), C15.0 LPC, C16.0 LPC, C16.0e LPC, C16.1 LPC, C16.1e LPC, C17.0 LPC, C18.0 LPC, C18.0e LPC, C18.1 LPC, C18.2 LPC, C20.0 LPC, C20.1 LPC, C20.3 LPC, C20.4 LPC, C22.6 LPC, C30.0 phosphatidylcholine (PC), C32.0 PC, C32.1 PC, C32.2 PC, C33.1 PC, C34.0 PC, C34.1 PC, C34.1e PC, C34.2 PC, C34.2e PC, C34.3e PC, C34.4PC, C35.1 PC, C35.2 PC, C36.1 PC, C36.2 PC, C36.2e PC, C36.3 PC, C36.4 PC, C36.4e PC, C36.5 PC, C36.5e PC, C37.4 PC, C38.3 PC, C38.4 PC, C38.4e PC, C38.5 PC, C38.6 PC, C40.4 PC, C40.4e PC, C40.5e PC, C40-.6 PC, C42.5e PC
Biomarkers of appetite/metabolomics (Method: LC; units: mM; part 2) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = Liquid Chromatography (LC); Units = mM; variables = C36.5 e Phosphatidyletjanolamine (PE), C38.5e PE, C38.6e PE, C32.1 Sphigomyelin (SM), C32.2 SM, C33.1 SM, C34.1 SM, C34.2 SM, C35.1 SM, C36.0 SM, C36.1 SM, C36.2 SM, C38.1 SM, C38.2 SM, C40.1 SM, C40.2 SM, C41.1 SM, C41.2 SM, C42.1 SM, C42.2 SM, C42.3 SM, C48.1 Triglyceride (TG), C48.2 TG, C50.1 TG, C50.2 TG, C50.3 TG, C50.4 TG, C51.2 TG, C52.1 TG, C52.2 TG, C52.3 TG, C52.4 TG, C52.5 TG, C54.2 TG, C54.3 TG, C54.4 TG, C54.5 TG
Biomarkers of appetite/metabolomics (Method: LC; units: ng/ml) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = Liquid Chromatography (LC); Units = ng/mL; variables = 5-hydroxytryptamine, 5-hydroxyindoleacetic acid, Trimethylamine-N-oxide
Biomarkers of appetite/metabolomics (Method: LC; units: uM; part 1) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = Liquid Chromatography (LC); Units = uM; variables = free carnitine, acetyl-carnitine, propionyl-carnitine, crotonyl-carnitine/methacrylyl-carnitine. isobutyryl-carnitine, butyryl-carnitink, hydroxybutyryl-carnitine a and b/3-hydroxyisobutyryl-carnitine, hydroxyvaleryl-carnitine, tiglyl-carnitine/3-methylcrotonyl-carnitine, 2-methyl-butyryl-carnitine, isovaleryl-carnitine/valeryl-carnitine, hexanoyl-carnitine, succinyl-carnitine, malonyl-carnitine
Biomarkers of appetite/metabolomics (Method: LC; units: uM; part 2) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = Liquid Chromatography (LC); Units = uM; variables = methyl-malonyl-carnitine, glutaryl-carnitine, adipyl-carnitine, octenoyl-carnitine, methylglutaryl-carnitine, octanoyl-carnitine, nonanoyl-carnitine, decadienoyl-carnitine, decenoyl-carnitine, decanoyl-carnitine/Fumaryl-carnitine, undecanoyl-carnitine, Glutaconyl-carnitine/iso-undecanoyl-carnitine, dodecenoyl-carnitine, dodecanoyl-carnitine, pimply-carnitine, tatradecadienyl-carnitine, tridecenoyl-carnitine, tatradecenoyl-carnitine, tatradecanoyl-carnitine, pentadecanoyl-carnitine/isopentadecanoyl-carnitine, hydroxyhexadecanoyl-carnitine a and b, hexadecadienyl-carnitine, octadecadienyl-carnitine, hexadecanoyl-carnitine, octadecenyl-carnitine, octadecanoyl-carnitine
Biomarkers of appetite/metabolomics (Method: GC; units: mM) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = Gas Chromatography (GC); Units = mM; variables = lactic acid, Glycolic acid, Alanine, Glycine, X2 Hydroxybutanoic acid, X3 Hydroxybutanoic acid, Valine, Leucine, Glycerol, Isoleucine, Proline, Gliceric acid, Serine, Threonine, Methionine, Ornithine, Glutamic acid, Phenylalanine, Lysine, Citric acid, Fructose, Glucose, Tyrosine, Palmatic acid, Linoleic acid, Oleic acid, Stearic acid, tryptophan, Sucrose, alpha-Tocopherol, Cholesterol
Biomarkers of appetite/metabolomics (Method: standard enzymatic methods; units: mg/dL) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = Standard enzymatic methods; Units = mg/dL; variables = v2 Glucose, v2 Cholesterol, v2 HDL cholesterol, v2 LDL cholesterol, v2 VLDL cholesterol, v2 triglyceride
Biomarkers of appetite/metabolomics (Method: standard enzymatic methods; units: U/L) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = Standard enzymatic methods; Units = U/L; variables = v2 Aspartate transaminase, v2 Alanine Transaminase, v2 Gamma glutamyl transferase,
Biomarkers of appetite/metabolomics (Method: standard enzymatic methods; units: mU/mL) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = Standard enzymatic methods; Units = mU/mL; variables = v2 insulin
Biomarkers of appetite/metabolomics (Method: MAGPIX; units: ug//mL) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = MAGPIX; Units = ug/mL; variables = v2 C-reactive protein, v2 Adiponectin
Biomarkers of appetite/metabolomics (Method: MAGPIX; units: ng//mL) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = MAGPIX; Units = ng/mL; variables = v2 Leptin
Biomarkers of appetite/metabolomics (Method: MAGPIX; units: pg//mL) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Willing participants will provide fasting blood samples and urine samples to allow for assessment of biomarkers of appetite and satiety which will be conducted.
  Method = MAGPIX; Units = pg/mL; variables = v2 Interleukin 6
Consumer benefits - Control of Eating Questionnaire (CoEQ) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  The CoEQ comprises 21-items that are designed to assess the severity and type of food cravings an individual experiences over the previous 24hrs or 7 days. Scores are presented using 100-mm visual analogue scales (VAS)
Consumer benefits - Three Factor Eating Questionnaire (TFEQ) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  The TFEQ comprises 51-items that are designed to assess three aspects of eating behaviour (restraint, 21 items; disinhibition, 16 items and hunger, 14 items). Each item scores 0 or 1 point. Individual subscale and total summed score will be analysed
Consumer benefits - Positive and Negative Affect Schedule (PANAS) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Comprises two 10 item mood scales, one that measures positive affect and the other which measures negative affect. Participants respond using 5-point scale that ranges from very slightly or not at all (1) to extremely (5).
Consumer benefits - Hospital Anxiety and Depression Scale (HADS) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Comprises 14 items designed to measure levels of anxiety (7 items) and depression (7 items). Each item on the questionnaire is scored from 0-3.
Consumer benefits - Dutch Eating Behaviour Questionnaire (DEBQ) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Comprises 33 items designed to measure three aspectings of eating behaviour (emotional eating, 13 items; external eating, 10 items and restrained eating, 10 items). Participants respond using 5-point scale that ranges from never (1) to very often (5). Higher scores indicate greater endorsement of that behaviour.
Consumer benefits - Power of Food Scale (PFS) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  The PFS comprises 15 items designed to assess the psychological impact of living in food-abundant environments. It measures appetite for, rather than consumption of, palatable foods, at three levels of food proximity (food available, food present, and food tasted). Participants respond using 5-point scale that ranges from Don't agree at all (1) to strongly agree (5).
Consumer benefits - Mindful Eating Scale (MES) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  The 29 item scale assesses the construct of mindul eating (a non-judgmental awareness of physical and emotional sensations associated with eating). Participants respond on a 4 point Likert scale (never, rarely, sometimes, usually)
Consumer benefits - Eating Self Efficacy Scale (ESES) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  The 25 item scale assesses eating when experiencing negative effect (15 items) and during socially accepted circumstances (10 items). Participants respond on a 7 point likert scale: no difficulty controlling eating (1) to most difficulty controlling eating (7).
Consumer benefits - Weight Self Efficacy Scale (WSES) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  The 20 item scale assesses confidence in managing eating (and subsequently keeping weight under control) in different situations. Responses are provided on a 9 point scale ranging from 0 = Not at all confident that you can resist the desire to eat to 9 = Very confident that you can resist the desire to eat.
Consumer benefits - Self Report Measure of Quality of Life (EQ-5D) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  This is a measure of health-related quality of life. It consists of a descriptive system and the EQ VAS. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. The scores on these five dimensions are converted to a single summary index number (utility).
Consumer benefits - Impact of Weight on Quality of Life-Lite (IWQOL) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  This is a 31-item, self-report, obesity-specific measure of health-related quality of life that consists of a total score and scores on each of five scales--physical function, self-esteem, sexual life, public distress, and work. Participants respond on a 5 point likert scale from never true (1) to always true (5)
Consumer benefits - Warwick Edinburgh Mental Well Being Scale (WEMWBS) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  WEMWBS is a 14 item scale with 5 response categories, summed to provide a single score ranging from 14-70. The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing.
Consumer benefits - Extended Satisfaction with Life Scale (ESWLS) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  The ESWLS is a 50-item self-report scale with responses rated on a seven point likert scale ranging from strongly agree to strongly disagree. Higher scores represent greater satisfaction. It measures satisfaction with life in nine domains (general life, social life, sexual life, relationships, self, physical appearance, family life, school life and job life). Scores for each subscale are calculated as the sum of the ratings for each of the items comprising the subscale.
Consumer benefits - Self-consciousness scale (SCSR) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  This is a 22 item scale with responses on a 4 point likert scale from 0 = "not like me at all" to 3 = "a lot like me". It comprises three dimensions: private self-consciousness, public self-consciousness and self anxiety. Scores for the subscales are calculated as the sum of the ratings for each of the items comprising the sub scale. The private self-consciousnes and social-anxiety sub scales contain items that are reverse coded.
Consumer benefits - Craving for Sweet Foods | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  This is a 6 item sub-scale of the Health and Taste Attitudes Questionnaire. Responses are provided on a 7 point likert scale from 1 = "strongly disagree" to 7 = "strongly agree". Responses predict well respondents self-reported consumption.
Consumer benefits - Perceived Stress Scale | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  This 10 item scale assesses an individual's feelings and thoughts over the last month. Items are designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. Responders select from 5 response options (0 = never; 4 = very often). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Consumer benefits - Pitsburg Sleep Quality Index | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. It contains both positively and negatively phrased items, with positively phrased items being reverse scored
Consumer benefits - International Physical Activity Questionnaire (IPAQ) | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  The International Physical Activity Questionnaires (IPAQ) assesses activity in 5 domains (job-related, transportation physical activity, at home, sport and leisure and time spent sitting) over the last seven days. It is self administered and provides a common instrument to obtain internationally comparable data on health-related physical activity.
Consumer benefits - Food Thought Suppression Inventory | Measured before the 8-week Low Calorie Diet period then after the 8-week Low Calorie Diet period and then after the 12-week intervention period
  Food Thought Suppression Inventory (FTSI) is a self-report measure. It contains 15- and 14-items, for women and men (regardless of BMI), respectively. Responses are provided on a 5 point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Scores can range from 15 to 75 with higher scores reflecting higher levels of food thought suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Halford, Professor, Principal Investigator — Univeristy of Liverpool
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No